CLINICAL TRIAL: NCT00622726
Title: Intravitreal Bevacizumab (AvastinTM) Injections Versus Conventional Laser Surgery for Vision-threatening Retinopathy of Prematurity: a Prospective, Randomized, Non-blinded, Controlled, Multi-center, Clinical Trial
Brief Title: Bevacizumab Eliminates the Angiogenic Threat for Retinopathy of Prematurity
Acronym: BEAT-ROP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Helen Mintz-Hittner, MD, Clinical Professor - Pediatric Ophthalmology, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-08-0036; IND: 101,578 (Other: Research to Prevent Blindness (NY, NY))
Record Dates: First submitted 2008-02-13; First posted 2008-02-25 (Estimated); Results first posted 2014-06-09 (Estimated); Last update posted 2017-06-06 (Actual); Status verified 2017-05

CONDITIONS: Retinopathy of Prematurity
Keywords: Vascular Endothelial Growth Factor; Angiogenesis Inhibitor; Premature infants; Bevacizumab; Zone I or Posterior Zone II ROP; Aggressive Posterior ROP; Stage 3 ROP; Neonatal Intensive Care Unit
MeSH Terms: conditions — Retinopathy of Prematurity; Premature Birth | interventions — Bevacizumab; Antibodies, Monoclonal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bevacizumab for ROP (Experimental): Intravitreal Bevacizumab Therapy is the Experimental Arm of this Study
  Interventions: Drug: Bevacizumab
- Conventional Laser for ROP (Active Comparator): Conventional Laser to the Peripheral Retina is the Control Arm of this Study
  Interventions: Procedure: Conventional Laser for ROP

INTERVENTIONS:
Drug: Bevacizumab — Anti-angiogenic drug: intravitreal injection of 0.625 mg (0.025 ml) once into each eye.
  Other Names: Avastin; Monoclonal antibody
  Arms: Bevacizumab for ROP
Procedure: Conventional Laser for ROP — Conventional Laser is applied to the Avascular Peripheral Retina (Anterior to the Vascularized Posterior Retina)
  Other Names: Diode Laser is the laser utilized for this study
  Arms: Conventional Laser for ROP

SUMMARY:
The purpose of this study was to determine the efficacy and additional advantages of intravitreal bevacizumab in the treatment of ROP for both Zone I and Zone II Posterior.

DETAILED DESCRIPTION:
This phase 2 study assessed the anti-neovascularization activity of intravitreal bevacizumab, as determined by regression of neovascular vessels of retinopathy of prematurity (ROP), in neonates with acute stage 3 ROP in zone I or posterior zone II with plus disease. This study enrolled 150 confirmed cases of vision threatening ROP which have definite plus disease [ranging from Early Treatment for Retinopathy of Prematurity, to Cryotherapy for Retinopathy of Prematurity . This was done because of the controversy regarding determining plus disease and the increasing concern that many infants are being treated whose ROP would spontaneously regress. Bevacizumab will be administered intravitreally using 0.625 mg (0.025 ml) injections into each eye. There was no intent to give additional doses unless there was a recurrence of vision threatening stage 3 ROP with plus disease since the disease is self limited by completion of vascularization. Clinical response and any evidence of ocular toxicities were documented by retinal imaging system (manufactured by Clarity Medical Systems, Inc.) taken pre-injection, one week and one month post injection, and at 6 months of age (54 weeks postmenstrual age)(window of 50 to 70 weeks PMA)(primary outcome) and at 12 months of age (80 weeks postmenstrual age)(window of 75 to 100 weeks PMA)(structural documentation). Using the same retinal imaging system, fluorescein angiograms have been taken when possible to document structural outcomes in greater detail. No evidence of systemic toxicities were documented by appropriate clinical and laboratory tests.

ELIGIBILITY:
Inclusion Criteria:

1. Infants who have been screened by the American Academy of Ophthalmology, the American Academy of Pediatrics, and the American Association for Pediatric Ophthalmology and Strabismus guidelines (≤1500 grams at birth and ≤30 weeks gestation) who develop Stage 3 ROP in zone I or posterior zone II.
2. Informed Consent from a parent or guardian.

Exclusion Criteria:

1. Infants who have a congenital systemic anomaly or have a congenital ocular abnormality.
2. Infants who cannot be treated by conventional laser therapy because of problems with media clarity. Generally, blind external cryotherapy would be utilized as an initial therapy and the infant would be excluded from the study even if the media clear subsequently.
3. Informed Consent from a parent or guardian refused. This will mean that an infant automatically will receive laser therapy. Bevacizumab (Avastin®) treatment cannot be given outside of the Protocol. No data will be used from an infant without Informed Consent.

Ages: 4 Weeks to 22 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2008-03 (Actual); Primary Completion 2010-08 (Actual); Study Completion 2020-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Helen A. Mintz-Hittner, M.D., Principal Investigator — The University of Texas Health Science Center, Houston
Locations (15):
- United States (15):
  - Huntington Memorial Hospital, Pasadena, California
  - Presbyterian-St. Luke's Hospital, Denver, Colorado
  - OSF St. Francis Medical Center-Children's Hospital of Illinois, Peoria, Illinois
  - Palmetto Health Richland Hospital, Columbia, South Carolina
  - Palmetto Health Baptist Hospital, Columbia, South Carolina
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Baylor University Medical Center, Dallas, Texas
  - Las Palmas Medical Center, El Paso, Texas
  - R.E. Thomason Hospital, El Paso, Texas
  - Del Sol Medical Center, El Paso, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - St. Joseph Medical Center, Houston, Texas
  - Children's Memorial Hermann Hospital, Houston, Texas
  - Memorial Hermann Southwest Hospital, Houston, Texas
  - Clear Lake Regional Medical Center, Webster, Texas

REFERENCES:
- [Background] Mintz-Hittner HA, Best LM. Antivascular endothelial growth factor for retinopathy of prematurity. Curr Opin Pediatr. 2009 Apr;21(2):182-7. doi: 10.1097/MOP.0b013e32832925f9. PMID 19300261
- [Background] Mintz-Hittner HA. Avastin as monotherapy for retinopathy of prematurity. J AAPOS. 2010 Feb;14(1):2-3. doi: 10.1016/j.jaapos.2009.12.002. No abstract available. PMID 20227612
- [Background] Mintz-Hittner HA. Intravitreal pegaptanib as adjunctive treatment for stage 3+ ROP shown to be effective in a prospective, randomized, controlled multicenter clinical trial. Eur J Ophthalmol. 2012 Sep-Oct;22(5):685-6. doi: 10.5301/ejo.5000176. PMID 22669847
- [Background] Mintz-Hittner HA. Treatment of retinopathy of prematurity with vascular endothelial growth factor inhibitors. Early Hum Dev. 2012 Dec;88(12):937-41. doi: 10.1016/j.earlhumdev.2012.09.019. Epub 2012 Oct 15. PMID 23078830
- [Result] Mintz-Hittner HA, Kuffel RR Jr. Intravitreal injection of bevacizumab (avastin) for treatment of stage 3 retinopathy of prematurity in zone I or posterior zone II. Retina. 2008 Jun;28(6):831-8. doi: 10.1097/IAE.0b013e318177f934. PMID 18536599
- [Result] Kong L, Mintz-Hittner HA, Penland RL, Kretzer FL, Chevez-Barrios P. Intravitreous bevacizumab as anti-vascular endothelial growth factor therapy for retinopathy of prematurity: a morphologic study. Arch Ophthalmol. 2008 Aug;126(8):1161-3. doi: 10.1001/archophthalmol.2008.1. No abstract available. PMID 18695118
- [Result] Mintz-Hittner HA, Kennedy KA, Chuang AZ; BEAT-ROP Cooperative Group. Efficacy of intravitreal bevacizumab for stage 3+ retinopathy of prematurity. N Engl J Med. 2011 Feb 17;364(7):603-15. doi: 10.1056/NEJMoa1007374. PMID 21323540
- [Result] Geloneck MM, Chuang AZ, Clark WL, Hunt MG, Norman AA, Packwood EA, Tawansy KA, Mintz-Hittner HA; BEAT-ROP Cooperative Group. Refractive outcomes following bevacizumab monotherapy compared with conventional laser treatment: a randomized clinical trial. JAMA Ophthalmol. 2014 Nov;132(11):1327-33. doi: 10.1001/jamaophthalmol.2014.2772. PMID 25103848
- [Result] Mintz-Hittner HA, Geloneck MM, Chuang AZ. Clinical Management of Recurrent Retinopathy of Prematurity after Intravitreal Bevacizumab Monotherapy. Ophthalmology. 2016 Sep;123(9):1845-55. doi: 10.1016/j.ophtha.2016.04.028. Epub 2016 May 27. PMID 27241619

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of recruitment: March 13, 2008 to August 4, 2010. Patients recruited were all in neonatal intensive care units.
Groups:
- Bevacizumab for ROP-Experimental Arm: Intravitreal Bevacizumab Therapy is the Experimental Arm of this Study. 31 patients had zone I ROP; 39 patients had zone II posterior ROP.
- Conventional Laser for ROP-Control Arm: Conventional Laser to the Peripheral Retina is the Control Arm of this Study. 33 patients had zone I ROP; 40 patients had posterior zone II ROP.
Period: March, 2008 to August, 2010
Arm/Group | Bevacizumab for ROP-Experimental Arm | Conventional Laser for ROP-Control Arm
Started | 75 | 75
Completed | 70 (All infants were extremely immature with multiple neonatal intensive care unit complications.) | 73 (All infants were extremely immature with multiple neonatal intensive care unit complications.)
Not Completed | 5 | 2
Not completed — Death | 5 | 2
Period: August, 2010 to April, 2013
Arm/Group | Bevacizumab for ROP-Experimental Arm | Conventional Laser for ROP-Control Arm
Started | 70 | 73
Completed | 69 | 68
Not Completed | 1 | 5
Not completed — Death | 1 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bevacizumab for ROP-Experimental Arm | Conventional Laser for ROP-Control Arm | Total
Number analyzed (Participants) | 75 | 75 | 150
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 75 | 75 | 150
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 0.2 (0.1) | 0.2 (0.1) | 0.2 (0.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 23 | 49
  Male | 49 | 52 | 101
Region of Enrollment [Number; unit: participants]
  United States | 75 | 75 | 150

OUTCOME MEASURES:

1. Primary Outcome: Number of Eyes Showing Recurrence of Neovascularization Arising From the Retinal Vessels and Requiring Re-treatment
Description: For Bevacizumab: Regrowth of new vessels at the site of the original extraretinal fibrovascular proliferation and/or at the site of the anterior edge of inner retinal vascularization.
  For Laser: Regrowth of new vessels from the vessels at the anterior edge of inner retinal vascularization (remaining after retinal ablation).
Time Frame: 54 weeks postmenstrual age (window of 50 to 70 weeks)
Population: Both eyes of all surviving infants were analyzed for recurrence: thus, 143 surviving infants and 286 eyes were analyzed. Reporting the number of eyes that developed recurrences
Measure: Number; unit: eyes with recurrences
Units Other Than Participants: Eyes
Groups:
- Bevacizumab for ROP-Experimental Arm: Intravitreal Bevacizumab Therapy is the Experimental Arm of this Study. 31 patients/62 eyes had zone I ROP; 39 patients/78 eyes had zone II posterior ROP.
- Conventional Laser for ROP-Control Arm: Conventional Laser to the Peripheral Retina is the Control Arm of this Study. 33 patients/66 eyes had zone I ROP; 40 patients/80 eyes had posterior zone II ROP.
Arm/Group | Bevacizumab for ROP-Experimental Arm | Conventional Laser for ROP-Control Arm
Number analyzed (Participants) | 70 | 73
Number analyzed (Eyes) | 140 | 146
eyes with recurrences | 6 | 32

2. Secondary Outcome: Myopia in Zone I and Posterior Zone II of Infant Eyes
Description: Myopia was determined via refraction using a retinoscope and lenses. Myopia is defined as a refractive error reported in Diopters.
Time Frame: 2.5 years of age
Population: As of 6/2013, there were 13 deaths/ 26 eyes. Exclusions from surviving 137 infants/ 274 eyes: 6 infants/19 eyes with intraocular surgery--leaving: 131 infants/ 255 eyes; 14 infants/ 21 eyes had recurrence and 22 infants/ 44 eyes were lost to follow-up--leaving: 95 infants/ 190 eyes. Thus, only the refractions on these infants/ eyes are given.
Measure: Mean (Standard Deviation); unit: Diopters
Units Other Than Participants: Eyes
Groups:
- Bevacizumab-Experimental Group: Zone I: The eyes of all surviving infants without recurrences and without any previous intra-ocular surgery who received bevacizumab will be examined: Zone I.
- Conventional Laser-Control Group: Zone I: The eyes of all surviving infants without recurrences and without any previous intra-ocular surgery who received conventional laser will be examined: Zone I.
- Bevacizumab Experimental Group: Posterior Zone II: The eyes of all surviving infants without recurrences and without any previous intra-ocular surgery who received bevacizumab will be examined: Posterior Zone II.
- Conventional Laser-Control Group: Posterior Zone II: The eyes of all surviving infants without recurrences and without any previous intra-ocular surgery who received conventional laser will be examined: Posterior Zone II.
Arm/Group | Bevacizumab-Experimental Group: Zone I | Conventional Laser-Control Group: Zone I | Bevacizumab Experimental Group: Posterior Zone II | Conventional Laser-Control Group: Posterior Zone II
Number analyzed (Participants) | 25 | 12 | 28 | 30
Number analyzed (Eyes) | 50 | 26 | 56 | 58
Diopters | -1.36 (3.34) | -7.34 (7.44) | -0.63 (2.56) | -5.20 (5.77)

3. Secondary Outcome: Visual Acuity
Description: The visual acuity will be measured at 20 feet with figures or letters from all infants able to cooperate.
Time Frame: Age 7 years.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: March, 2008 to April 2013
Description: No adverse events have occurred (with the exception of 6 deaths in the bevacizumab arm and 7 deaths in the conventional laser arm.
Arm/Group | Bevacizumab for ROP-Experimental Arm | Conventional Laser for ROP-Control Arm
Serious Adverse Events (participants affected / at risk) | 0/69 | 0/68
Other Adverse Events (participants affected / at risk) | 0/69 | 0/68

LIMITATIONS AND CAVEATS:
Limitations:

1. number of patients is too small to determine efficacy of bevacizumab in posterior zone II ROP.
2. number of patients is too small to determine safety of bevacizumab systemically.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No